CLINICAL TRIAL: NCT03708432
Title: An Observational, Retrospective Study of 500mg Fulvestrant in Hormone Receptor+/HER2- Advanced Breast Cancer
Brief Title: 500mg Fulvestrant in HR+ MBC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-4
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fulvestrant: Fulvestrant 500mg per month (D1, D28, q28d), with a loading dose 500mg of first dose at D15

SUMMARY:
To study the real world use of 500mg Fulvestrant in HR+ MBC.

DETAILED DESCRIPTION:
An observational, retrospective study of 500mg Fulvestrant in hormone receptor+/HER2- advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ER/PR+，HER2- advanced breast cancer
2. Advanced breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.

3.500mg Fulvestrant treatment of advanced breast cancer for at least one month, between Jan 2011 and Dec 2015.

4.Available medical history

Exclusion Criteria:

1. Incomplete medical history
2. HER2 overexpression or gene amplification, ie, immunohistochemistry (IHC) 3+ or fluorescence in situ hybridisation (FISH)+, where appropriate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao Y, Li Y, Gong C, Xie Y, Zhang J, Wang L, Cao J, Tao Z, Wang B, Hu X. Optimal duration of prior endocrine therapy predicts the efficacy of Fulvestrant in a real-world study for patients with hormone receptor-positive and HER2-negative advanced breast cancer. Cancer Med. 2020 Dec;9(23):8821-8831. doi: 10.1002/cam4.3491. Epub 2020 Oct 6. PMID 33022852